CLINICAL TRIAL: NCT01564992
Title: Drug Interaction With Genes in Parkinson's Disease
Acronym: DIGPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P 071240
Record Dates: First submitted 2012-02-23; First posted 2012-03-28 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Pharmacogenetics; Genetics
MeSH Terms: conditions — Parkinson Disease | interventions — Polymorphism, Genetic; Haplotypes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson disease: Identification of genes
  Interventions: Other: Identification of genes

INTERVENTIONS:
Other: Identification of genes — Identification of genes which polymorphism or haplotype is associated with a complication of Parkinson disease, directly or with the interaction of treatment.
  Other Names: polymorphism or haplotype

SUMMARY:
This observational study aims at identifying gene modifiers of Parkinson Disease (PD) and of treatment response and adverse events of antiparkinsonian drugs. Six hundred PD patients will be followed annually for up to 5 years. A biological collection will be associated with a full clinical assessment of motor and non motor symptoms, medical and treatment history, environmental factors. The association between candidate gene polymorphisms and disease or treatment complications will be analyzed.

DETAILED DESCRIPTION:
Title : Drug interaction with genes in Parkinson Disease

Objective:

To identify genes associated to disease and treatment complication and response.

Number of subjects: 500

Study duration : 6 years

Design:

Prospective cohort with biological collection

Primary objective:

Identification of genes which polymorphism or haplotype is associated with a complication of Parkinson disease, directly or with the interaction of treatment.

Secondary objectives:

* Prevalence and incidence of disease or treatment complications
* Clinical risk factor for disease or treatment complications
* Biomarkers of disease progression, disease or treatment complications

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age > 18.
* Parkinson Disease according to UKPDSBB criteria
* PD diagnosis < 6 years
* Informed consent

Exclusion Criteria:

- Atypical parkinsonism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women adults with a Parkinson Disease according to UKPDSBB criteria, diagnosed < 6 years
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-05 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
All complications of the disease or treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Corvol, MD, PhD, Principal Investigator — Asssitance Publique - Hopitaux de Paris
Locations (1):
- Centre d'Investigation Clinique Neuro - Bâtiment ICM - Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marques A, Vidal T, Pereira B, Benchetrit E, Socha J, Pineau F, Elbaz A, Artaud F, Mangone G, You H, Cormier F, Galitstky M, Pomies E, Rascol O, Derkinderen P, Weintraub D, Corvol JC, Durif F; DIGPD study group. French validation of the questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS). Parkinsonism Relat Disord. 2019 Jun;63:117-123. doi: 10.1016/j.parkreldis.2019.02.026. Epub 2019 Mar 4. PMID 30862454
- [Derived] Corvol JC, Artaud F, Cormier-Dequaire F, Rascol O, Durif F, Derkinderen P, Marques AR, Bourdain F, Brandel JP, Pico F, Lacomblez L, Bonnet C, Brefel-Courbon C, Ory-Magne F, Grabli D, Klebe S, Mangone G, You H, Mesnage V, Lee PC, Brice A, Vidailhet M, Elbaz A; DIGPD Study Group. Longitudinal analysis of impulse control disorders in Parkinson disease. Neurology. 2018 Jul 17;91(3):e189-e201. doi: 10.1212/WNL.0000000000005816. Epub 2018 Jun 20. PMID 29925549